CLINICAL TRIAL: NCT05847322
Title: A Human Controlled Infection Study to Establish Safety of Infection With Bordetella Pertussis With Antibiotic Therapy Delayed for up to 6 Weeks
Brief Title: Periscope Phase C Bordetella Pertussis Human Challenge Study With Delayed Antibiotic Therapy for 6 Weeks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRAS 304211; 68737 (Other: ERGO)
Record Dates: First submitted 2023-03-07; First posted 2023-05-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Pertussis/Whooping Cough
MeSH Terms: conditions — Whooping Cough | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Single centre controlled human Bordetella pertussis colonisation study. Intervention: nasal challenge with Bordetella pertussis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contact (Other): Contact volunteers are those volunteers whose partner/spouse is a Challenge volunteer. Investigators will monitor Contact volunteers to collect information about transmission. A 3 day course of Azithromycin will be administered on week 6 if colonised.
  Interventions: Drug: Azithromycin Pill
- Challenge (Experimental): Challenge volunteers will receive a nasal inoculation containing Bordetella pertussis on Day 0. They will return to the Clinical Research Facility weekly to monitor safety, colonisation and immune responses. A 3 day course of Azithromycin will be administered on week 6 if colonised.
  Interventions: Biological: Bordetella pertussis B1917; Drug: Azithromycin Pill

INTERVENTIONS:
Biological: Bordetella pertussis B1917 — The B. pertussis isolate to be used in this human colonisation model is strain B1917, which is representative of current isolates in Europe. The strain, isolated in 2000 from a Dutch patient with B. pertussis disease, expresses Pertactin (PRN), Pertussis Toxin (PT) and Filamentous Haemagglutinin (FHA). This strain has been extensively characterised in the mouse model as well as by proteomics and transcriptomics and has a closed genome available. It is fully sensitive to azithromycin in vitro.
  Arms: Challenge
Drug: Azithromycin Pill — A 3 day course of azithromycin will be administered to all colonised volunteers at week 6, or sooner if early pertussis disease is suspected

SUMMARY:
Primary objective- To assess the safety of nasal inoculation of healthy volunteers with B. pertussis with antibiotic therapy given to eradicate colonisation at 6 weeks after inoculation or at symptom onset, whichever occurs first

Secondary objectives - To measure the rate of natural clearance of carriage of B. pertussis following nasal inoculation

* To assess the kinetics of B. pertussis colonisation density following nasal inoculation
* To describe the microevolution of B. pertussis and adaptation of the resident microbiome during B. pertussis carriage
* To measure B. pertussis-specific antibody and cellular immunological responses in healthy volunteers during colonisation with B. pertussis - To identify biomarkers that correlate with natural clearance of B. pertussis carriage after induced B. pertussis colonisation
* To detect transmission of B. pertussis to bedroom contacts of inoculated volunteers during prolonged asymptomatic colonisation

DETAILED DESCRIPTION:
This is a prospective controlled human challenge study; Challenge group: The challenge volunteers will be healthy volunteers, aged 18-55 years, not having close contact with people having increased risk of severe pertussis complications or increased risk of transmitting to vulnerable individuals. Eligible volunteers must be willing to abide by infection control measures during social contact and to attend immediately if they become symptomatic. People who live in institutions in which multiple people share dormitory facilities, such as boarding schools or military barracks will be excluded.

The standard inoculum, a dose of 105 cfu, determined in Phase A of the Bp human challenge study, will be used. Participants will be followed up weekly and colonisation will be measured in nasal washes. If culture of the nasal wash taken at week 5 following nasal inoculation is positive for B. pertussis, then eradication therapy will be given at week 6. Early eradication therapy will be given if a participant presents with symptoms of early B. pertussis disease.

Recruitment will continue until 10 challenge volunteers have been colonised and then completed study participation to week 6 as per protocol. Volunteers who withdraw from the study early or have colonisation cleared with antibiotic treatment given for any reason will be replaced. Assuming a colonisation fraction of at least 30% and allowing for study withdrawal the investigator expect a maximum number of 36 volunteers to be inoculated.

Contact group: A group of contact volunteers, maximum 36 individuals, will be enrolled to assess transmission by monitoring for colonisation with the challenge strain of B. pertussis. These contact volunteers will be bedroom sharers of challenge volunteers and will give informed consent for their participation in the study, prior to inoculation of the corresponding challenge volunteer. Eradication therapy will be given at week 6 if the culture of nasal wash is positive for B. pertussis at week 5. Early eradication therapy will be given if a contact volunteer presents with symptoms of early B. pertussis disease.

Challenge and contact volunteers will be required to agree to infection control measures prior to enrolment in the study. Part of this agreement will be to refrain from bedroom sharing or intimate contact with any individual other than one declared and consented bedroom contact. They will avoid contact with children or people vulnerable to whooping cough such as unimmunised or partially immunised children and infants aged < 1 year, and pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 55 years inclusive on the day of screening
* Fully conversant in the English language
* Able to communicate easily by both mobile telephone, email and text messaging
* Able and willing (in the investigator's opinion) to comply with all study requirements
* Written informed consent to participate in the study
* Willingness to take a curative antibiotic regimen if / when required according to the study protocol
* Willingness to abide by infection control guidelines during social contact for the duration of their participation in the study
* Willingness to attend to the National Institute for Health Research (NIHR) Clinical Research Facility (CRF) Southampton immediately if they become symptomatic
* Agreement to have no bedroom contacts other than their corresponding contact/challenge volunteer between inoculation and 6 weeks after inoculation
* Able to answer all questions on the pre-consent questionnaire correctly

Exclusion Criteria:

* Individuals living in the same households as:

  1. unimmunised or partially immunised children and infants aged < 1 year
  2. pregnant women >32 weeks who have not received pertussis vaccination at least a week prior to contact
  3. immunosuppressed individuals
  4. frail individuals
  5. healthcare workers regularly working with vulnerable individuals as above
* Individuals who have inviolable commitments within the study period (from day 0 to week 6 + 2 days) to be in close contact with:

  1. unimmunised or partially immunised children and infants aged < 1 year
  2. pregnant women >32 weeks who have not received pertussis vaccination at least a week prior to contact
  3. immunosuppressed individuals
  4. frail individuals
* Individuals who live in a boarding school or dormitory during the study.
* B. pertussis detected on nasal wash taken before the initial challenge
* Individuals with a confirmed or suspected infection at the time of inoculation with B. pertussis
* Individuals who have participated in other interventional clinical trials in the last 12 weeks
* Individuals who have a history of receiving B. pertussis vaccination in the last 5 years
* Individuals who have previously participated in a B. pertussis human challenge study
* Individuals who have had a proven B. pertussis infection in the last 5 years
* Individuals who have a history of never being vaccinated against B. pertussis
* Current smokers defined as having had a cigarette/cigar in the last week (including vaping)
* Use of systemic antibiotics within 30 days of or during the challenge
* Any confirmed or suspected immunosuppressive or immune-deficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (topical steroids are allowed)
* Use of immunoglobulins or blood products within 3 months prior to enrolment
* History of allergic disease or reactions likely to be exacerbated by any component of the inoculum
* Contraindications to the use of azithromycin or macrolides
* Pregnancy, lactation or intention to become pregnant during the study
* Any clinically significant abnormal finding on biochemistry, haematology, toxicology or serological blood tests, urinalysis (see The following reference ranges are provided for the purpose of guidance only. Results that fall outside of these ranges may not be of clinical significance but should be considered on an individual basis.) or clinical examination - in the event of abnormal test results, confirmatory repeat tests will be requested
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data, for example recent surgery to the nasopharynx

Exclusion criteria - Contact volunteers

* Individuals living in the same households as:

  1. unimmunised or partially immunised children and infants aged < 1 year
  2. pregnant women
  3. immunosuppressed individuals
  4. frail individuals
  5. healthcare workers working with vulnerable individuals as above
* Individuals who have inviolable commitments within the study period (from day 0 to week 6 + 2 days) to be in close contact with:

  1. unimmunised or partially immunised children and infants aged < 1 year
  2. pregnant women >32 weeks who have not received pertussis vaccination at least a week prior to contact
  3. immunosuppressed individuals
  4. frail individuals
* Individuals who have been involved in other clinical trials involving receipt of an investigational product over the last 12 weeks or if there is planned use of an investigational product during the study period
* Individuals who have previously participated in a B. pertussis human challenge study
* Individuals who have a history of never being vaccinated against B. pertussis
* Any confirmed or suspected immunosuppressive or immune-deficient state, including HIV infection; malignancy, asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (topical steroids are allowed)
* Contraindications to the use of azithromycin or macrolides
* Any clinically significant abnormal finding on clinical examination
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Pregnancy, lactation or intention to become pregnant during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To assess the incidence of solicited adverse events during prolonged colonisation with Bordetella pertussis following nasal inoculation of healthy adult volunteers | 6 weeks.
  • Participants will be asked about the occurrence of solicited adverse events at standardised visits. Any symptoms will be recorded and assessed by a study doctor. If deemed necessary by the study doctor further tests will be requested
To assess the incidence of unsolicited adverse events during prolonged colonisation with Bordetella pertussis following nasal inoculation of healthy adult volunteers | 6 weeks.
  Participants will be asked about the occurrence of unsolicited adverse events at standardised visits. Any symptoms will be recorded and assessed by a study doctor. If deemed necessary by the study doctor further tests will be requested
To establish the rate of natural clearance of Bordetella pertussis colonisation as detected by nasal wash. | 6 weeks.
  Bordetella pertussis colonisation will be measured weekly by culture of nasal washes. Putative positive cultures will be confirmed by polymerase chain reaction (PCR).
To establish the rate of natural clearance of Bordetella pertussis colonisation as detected by nasopharyngeal swab | 6 weeks.
  Bordetella pertussis colonisation will be measured weekly by culture of nasopharyngeal swabs. Putative positive cultures will be confirmed by polymerase chain reaction (PCR).

SECONDARY OUTCOMES:
To establish the change in colonisation density of Bordetella pertussis during prolonged colonisation as measured from nasal wash samples | 6 weeks.
  Bordetella pertussis colonisation density will be measured weekly by culture of nasal washes. Putative positive cultures will be confirmed by polymerase chain reaction (PCR).
To establish the change in colonisation density of Bordetella pertussis during prolonged colonisation as measured by nasopharyngeal swab samples | 6 weeks.
  Bordetella pertussis colonisation density will be measured weekly by culture of nasopharyngeal swabs. Putative positive cultures will be confirmed by polymerase chain reaction (PCR).
To establish the occurrence of transmission to close contacts during prolonged Bordetella pertussis colonisation | 6 weeks.
  Bordetella pertussis colonisation density will be measured weekly by culture of nasal washes. Putative positive cultures will be confirmed by polymerase chain reaction (PCR).
To establish any association between baseline anti-PT IgG level and protection from colonisation with Bordetella pertussis | Day 0
  Anti-PT IgG will be measured in blood at baseline (Day 0)
To establish any association between baseline anti-PRN IgG level and protection from colonisation with Bordetella pertussis | Day 0
  Anti-PRN IgG will be measured in blood at baseline (Day 0)
To establish any association between baseline anti-FHA IgG level and protection from colonisation with Bordetella pertussis | Day 0
  Anti-FHA IgG will be measured in blood at baseline (Day 0)
To establish any association between baseline anti-FIM IgG level and protection from colonisation with Bordetella pertussis | Day 0
  Anti-FIM IgG will be measured in blood at baseline (Day 0)
To monitor change in anti-PT IgG levels during prolonged colonisation with Bordetella pertussis | 6 weeks.
  Anti-PT IgG will be measured in blood at standardised timepoints
To monitor change in anti-PRN IgG levels during prolonged colonisation with Bordetella pertussis | 6 weeks.
  Anti-PRN IgG will be measured in blood at standardised timepoints
To monitor change in anti-FHA IgG levels during prolonged colonisation with Bordetella pertussis | 6 weeks.
  Anti-FHA IgG will be measured in blood at standardised timepoints
To monitor change in anti-FIM IgG levels during prolonged colonisation with Bordetella pertussis | 6 weeks.
  Anti-FIM IgG will be measured in blood at standardised timepoints
To monitor change in anti-PT IgG levels associated with natural clearance of Bordetella pertussis | 6 weeks.
  Anti-PT IgG will be measured in blood at standardised timepoints
To monitor change in anti-PRN IgG levels associated with natural clearance of Bordetella pertussis | 6 weeks.
  Anti-PRN IgG will be measured in blood at standardised timepoints
To monitor change in anti-FHA IgG levels associated with natural clearance of Bordetella pertussis | 6 weeks.
  Anti-FHA IgG will be measured in blood at standardised timepoints
To monitor change in anti-FIM IgG levels associated with natural clearance of Bordetella pertussis | 6 weeks.
  Anti-FIM IgG will be measured in blood at standardised timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- NIHR Clinical Research Facility, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No